CLINICAL TRIAL: NCT06116903
Title: Clinical Relevance of Detecting Molecular Abnormalities in Glial Tumor Exosomes
Acronym: ExoGLIE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI22_0011-ExoGLIE
Record Dates: First submitted 2023-10-31; First posted 2023-11-03 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Detection of molecular abnormalities (Experimental): Blood samples will be taken from 2 + 3 Cell-Free DNA Collection tubes (Roche): for the comparative performance of the two methods (main objective) 3 Cell-Free DNA Collection tubes will be collected at 3 months (post chemotherapy) to evaluate the clinical relevance of a new analysis of molecular alterations on exosomes
  Interventions: Genetic: Blood sampling

INTERVENTIONS:
Genetic: Blood sampling — Blood sampling for testing of the detection of molecular abnormalities in exosomes of glial tumors

SUMMARY:
The purpose of this pilot study is that exosomes constitute a more interesting support for analyzes allowing a broader screening of molecular alterations to be carried out with more reliable, more sensitive and more efficient results than the reference Foundation One Liquid CDx test.

DETAILED DESCRIPTION:
Gliomas are the most common primary brain tumors in adults. The heterogeneity of tumors, the lack of reliable criteria for identifying different subtypes make their histopathological diagnosis and their management complex. The molecular profiling from circulating exosomes is one of the most promising approaches to better characterize gliomas.

We will demonstrate the superiority of detection by NGS of molecular abnormalities present in exosomes from glioblastomas, compared to detection by the Foundation One Liquid CDx test on ctDNA.

ELIGIBILITY:
Inclusion Criteria:

* Subject of both sexes at least 18 years of age with glioblastoma.
* Patient for whom an FMI test is indicated, progressing after a 1st line following the chemotherapy and radiotherapy protocol (STUPP protocol)
* Patient affiliated to French social security

Exclusion Criteria:

* Patient included in another research protocol using an experimental molecule.
* Any medical or psychiatric condition which, in the Investigator's opinion, would preclude the patient from adhering to the protocol or completing the study per protocol
* Patient under legal protection, guardianship or curatorship
* Patient with active malignancy or a previous malignancy within the past 5 years; except for patient with resected Basocarcinoma and resected carcinoma in-situ of the cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Analyse Next-generation sequencing (NGS) | 3 months
  Higher proportion of contributory samples identified by NGS analysis (via exosomes) compared to that of FMI (Foundation Medicine International) test (at inclusion)

SECONDARY OUTCOMES:
Expression of biomarkers | 3 months
  Level of expression of biomarkers, for the same patient, by molecular analysis of exosomes and blood sampling according to the FMI test protocol
Molecular alterations | 3 months
  Modification or not modification of the profile of the molecular alterations
carbon footprint | 3 months
  Evaluation of the carbon footprint for each of the 2 techniques (NGS via exosomes and FMI test)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No